CLINICAL TRIAL: NCT03510936
Title: Effect of Probiotics on the Gut Mircobiome of Infants With Jaundice
Brief Title: Gut Microbiome Associated Study of Shanghai Infants With Jaundice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Director, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHSYEK2018
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Gastrointestinal Microbiome
Keywords: Probiotics; Gut Microbiome; Infants; Jaundice
MeSH Terms: conditions — Jaundice | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blue light phototherapy (No Intervention): the patients in this arm will not receive probiotics.
- probiotics concurrent with phototherapy (Experimental): the patients in this arm will receive probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus, Enterococcus faecalis for 2 weeks
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — the patients in this arm will receive probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus, Enterococcus faecalis with does of 1.5*10^7CFU for 2 weeks
  Arms: probiotics concurrent with phototherapy

SUMMARY:
The purpose of this study is to evaluate the effect of probiotics on the gut microbiome of infants with jaundice.

DETAILED DESCRIPTION:
This study aims to examin the impact of probiotics administration during the process of infants jaundice treatment and recovery phase.the recovery phase.Birth,7 days,14 days and 42 days data will be collected and put into analysis to provide some suggestions on the probiotics use in the clinical for the infants with jaundice.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with jaundice treated with blue light phototherapy

Exclusion Criteria:

* Gestational weeks <37 Birth weight <2500g or ≥4000g History of asphyxia anoxia at birth With infectious diseases treated with antibiotic With congenital metabolic diseases or hereditary diseases With gastrointestinal diseases

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
change from birth,7 days,14 days on gut microbiome at 42 days by 16S rRNA | 42 days
  change of the gut microbiome will be calculated at 42 days in comparison with birth,7 days,14 days

SECONDARY OUTCOMES:
change from birth on gut microbiome at 7 days by 16S rRNA | 7 days
  change of the gut microbiome will be calculated at 7 days in comparison with baseline
change from birth and 7 days on gut microbiome at 14 days by 16S rRNA | 14 days
  change of the gut microbiome will be calculated at 14 days in comparison with birth and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Huanlong Qin, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, China